CLINICAL TRIAL: NCT02344030
Title: Comparative Study of King Vision® Standard Blade and King Vision® Channeled for Tracheal Intubation: a Prospective Randomised Study
Brief Title: Comparsion of King Vision® Standard Blade and King Vision® Channeled Blade in Patients Scheduled for Tracheal Intubation
Acronym: KingVision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Marc Kriege, MD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGUKV
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Hypoxemia
Keywords: airway; videolaryngoscope
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard blade (Experimental): Standard Blade: tracheal intubation with standard blade
  Interventions: Device: channeled blade; Device: standard blade
- channeled blade (Experimental): Channeled Blade: tracheal intubation with channeled blade
  Interventions: Device: channeled blade; Device: standard blade

INTERVENTIONS:
Device: channeled blade — In a randomised trial we measure the time for ventilation by means of endtidale CO2 Curve
Device: standard blade — In a randomised trial we measure the time for ventilation by means of endtidale CO2 Curve

SUMMARY:
Comparison of intubation time from the time to fix the Trachealtube to the first end-tidal CO2 ventilation by means of the curve on the ventilator at KV standard blade and KV channeled blade

DETAILED DESCRIPTION:
In the proposed clinical trial the time measured until the first manual ventilation at 44 study participants with elective anesthesia by using the KV standard blade and KV channeled blade. Bedside the time for tracheal intubation, we documented the view on the monitor which is connected to the instrument, the C& L classification and POGO Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years No concurrent participation in another study
* capacity to consent
* Present written informed consent of the research participant
* Elective surgery under general anesthesia

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients
* Emergency situations in the context of a Difficult Airway Management
* ASA classification> 3
* situations where the possibility of accumulated gastric contents
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
comparison of different time for tracheal intubation | <2min
  We want to measure the time for tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Result] Murphy LD, Kovacs GJ, Reardon PM, Law JA. Comparison of the king vision video laryngoscope with the macintosh laryngoscope. J Emerg Med. 2014 Aug;47(2):239-46. doi: 10.1016/j.jemermed.2014.02.008. Epub 2014 Apr 16. PMID 24742495
- [Result] Akihisa Y, Maruyama K, Koyama Y, Yamada R, Ogura A, Andoh T. Comparison of intubation performance between the King Vision and Macintosh laryngoscopes in novice personnel: a randomized, crossover manikin study. J Anesth. 2014 Feb;28(1):51-7. doi: 10.1007/s00540-013-1666-9. Epub 2013 Jun 30. PMID 23812581
- [Derived] Kriege M, Alflen C, Noppens RR. Using King Vision video laryngoscope with a channeled blade prolongs time for tracheal intubation in different training levels, compared to non-channeled blade. PLoS One. 2017 Aug 31;12(8):e0183382. doi: 10.1371/journal.pone.0183382. eCollection 2017. PMID 28859114